CLINICAL TRIAL: NCT01485627
Title: Randomized Controlled Trial(RCT)of Patient, Caregiver and Physician Communication Coaching in Advanced Cancer
Brief Title: VOICE: Values and Options in Cancer Care
Acronym: VOICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ronald Epstein, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 35388; R01CA140419-01A2 (NIH)
Record Dates: First submitted 2011-11-30; First posted 2011-12-05 (Estimated); Results first posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Cancer
Keywords: Cancer; Communication; prognosis
MeSH Terms: conditions — Neoplasms; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Oncologists will receive communication training. Patients will be coached to make the most of the oncologist visit.
  Interventions: Behavioral: Communication training and coaching
- Control (No Intervention): Patients will receive usual care

INTERVENTIONS:
Behavioral: Communication training and coaching — Oncologists will receive communication training. Patients will be coached to make the most of the oncologist visit.
  Arms: Intervention

SUMMARY:
The purpose of this study is to determine whether a combined intervention for patients, caregivers and oncologists improves communication, quality of life, and quality of care.

DETAILED DESCRIPTION:
The purpose of this study is to (a) determine whether a combined intervention for patients, caregivers and physicians improves communication regarding treatment choices and prognosis in cancer, (b) to determine whether the intervention improves patient and caregiver well-being, quality of life and sense of peace, and (c) to determine whether the intervention affects health services utilization.

ELIGIBILITY:
Inclusion Criteria: Physicians

* Currently in clinical practice at participating institutions
* Oncologist that cares for patients with solid tumors
* Not planning to leave the practice during the next 6 months

Inclusion Criteria: Patients

* Currently a patient of an enrolled physician
* Age 21 years or older
* Diagnosis of advanced cancer
* Able to understand spoken English (study personnel will read materials to low literacy patients)

Inclusion Criteria: Caregivers

* Caregiver of a patient currently enrolled in the study
* Age 21 years or older
* Able to understand spoken English (study personnel will read materials to low literacy patients)

Exclusion Criteria: Physicians

* Non Physicians and physicians who are not oncologists
* Oncologists who exclusively care for patients with hematological malignancies
* Prior involvement in health-related coaching interventions

Exclusion Criteria: Patients

* Unable to complete orally-administered surveys in English
* Hospitalized or in hospice care at the time of recruitment
* Prior involvement in health-related coaching interventions
* Anticipating bone marrow transplantation or diagnosed with leukemia or lymphoma

Exclusion Criteria: Caregiver

Unable to complete orally-administered surveys in English

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Epstein, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Derived] Epstein RM, Duberstein PR, Fenton JJ, Fiscella K, Hoerger M, Tancredi DJ, Xing G, Gramling R, Mohile S, Franks P, Kaesberg P, Plumb S, Cipri CS, Street RL Jr, Shields CG, Back AL, Butow P, Walczak A, Tattersall M, Venuti A, Sullivan P, Robinson M, Hoh B, Lewis L, Kravitz RL. Effect of a Patient-Centered Communication Intervention on Oncologist-Patient Communication, Quality of Life, and Health Care Utilization in Advanced Cancer: The VOICE Randomized Clinical Trial. JAMA Oncol. 2017 Jan 1;3(1):92-100. doi: 10.1001/jamaoncol.2016.4373. PMID 27612178
- [Derived] Hoerger M, Epstein RM, Winters PC, Fiscella K, Duberstein PR, Gramling R, Butow PN, Mohile SG, Kaesberg PR, Tang W, Plumb S, Walczak A, Back AL, Tancredi D, Venuti A, Cipri C, Escalera G, Ferro C, Gaudion D, Hoh B, Leatherwood B, Lewis L, Robinson M, Sullivan P, Kravitz RL. Values and options in cancer care (VOICE): study design and rationale for a patient-centered communication and decision-making intervention for physicians, patients with advanced cancer, and their caregivers. BMC Cancer. 2013 Apr 9;13:188. doi: 10.1186/1471-2407-13-188. PMID 23570278

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 54 physicians were assessed for eligibility. Of these 2 were ineligible and 9 refused participation. 43 physicians were included in the pre-randomized phase and of these 2 withdrew and 3 did not enroll enough patients. Patients from 38 physicians were included for the cluster randomized clinical trial phase of the study.
Pre-assignment Details: 233 caregivers and 316 patients were consented. 204 caregivers were allocated and 127 of them were bereaved. 24 caregivers failed screening and 5 withdrew during screening. 26 patients failed screening and 9 withdrew during screening.
Units Other Than Participants: physicians
Groups:
- Intervention: Communication: Oncologists will receive communication training. Patients will be coached to make the most of the oncologist visit.
  Communication training and coaching: Oncologists will receive communication training. Patients will be coached to make the most of the oncologist visit.
- Control: Usual Care: Patients will receive usual care
Period: Overall Study
Arm/Group | Intervention: Communication | Control: Usual Care
Started | 244; 19 physicians (139 patients and 105 caregivers) | 241; 19 physicians (142 patients and 99 caregivers)
Allocated Caregivers: Total | 105; 19 physicians | 99; 19 physicians
Bereaved Caregivers: Total | 63; 19 physicians | 64; 19 physicians
Bereaved Caregivers: 1 Month | 51; 19 physicians | 51; 19 physicians
Bereaved Caregivers: 2 Month Completed | 49; 19 physicians | 52; 19 physicians
Bereaved Caregivers: 7 Month Completed | 48; 19 physicians | 49; 19 physicians
Completed | 178; 19 physicians (130 patients and 48 caregivers) | 184; 19 physicians (135 patients and 49 caregivers)
Not Completed | 66; 0 physicians | 57; 0 physicians
Not completed — Patient withdrew | 6 | 5
Not completed — Patient died | 3 | 1
Not completed — Patient lost to followup | 0 | 1
Not completed — Caregiver withdrew | 3 | 3
Not completed — Caregiver lost to follow up | 11 | 12
Not completed — Caregiver died | 1 | 0
Not completed — caregiver was not bereaved | 42 | 35

BASELINE CHARACTERISTICS:
Population: Patients: 130 for the intervention and 135 for the control arms, who completed the audio-recorded office visit. Caregivers: 50 for the intervention and 53 for the control arms, who were bereaved and completed the month 2 and/or month 7 assessment.
Groups:
- Intervention: Communication Training: Oncologists will receive communication training. Patients will be coached to make the most of the oncologist visit.
  Communication training and coaching: Oncologists will receive communication training. Patients will be coached to make the most of the oncologist visit.
- Total: Total of all reporting groups
Arm/Group | Intervention: Communication Training | Control: Usual Care | Total
Number analyzed (Participants) | 180 | 188 | 368
Age, Categorical [Count of Participants; unit: Participants] — Population: Age categorical was collected for the bereaved caregivers only who completed the month 2 and/or month 7 assessment.
  Participants
    number analyzed (Participants) | 50 | 53 | 103
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 21 | 27 | 48
    >=65 years | 29 | 26 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] — Continuous age was only collected for the patients. Categorical age was only collected for the caregivers. Population: Age continuous was collected for the patients.
  years
    number analyzed (Participants) | 130 | 135 | 265
    (all) | 64.2 (11.7) | 64.5 (11) | 64.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The overall number of participants is the total of caregivers and patients for each arm.
  Participants
    patients: number analyzed (Participants) | 130 | 135 | 265
    patients: Female | 76 | 70 | 146
    patients: Male | 54 | 65 | 119
    Caregivers: number analyzed (Participants) | 50 | 53 | 103
    Caregivers: Female | 25 | 29 | 54
    Caregivers: Male | 25 | 24 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Overall baseline participants includes both the patients and caregivers
  Participants
    patients: number analyzed (Participants) | 130 | 135 | 265
    patients: American Indian or Alaska Native | 0 | 0 | 0
    patients: Asian | 0 | 0 | 0
    patients: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    patients: Black or African American | 0 | 0 | 0
    patients: White | 116 | 119 | 235
    patients: More than one race | 0 | 0 | 0
    patients: Unknown or Not Reported | 14 | 16 | 30
    Caregivers: number analyzed (Participants) | 50 | 53 | 103
    Caregivers: American Indian or Alaska Native | 0 | 0 | 0
    Caregivers: Asian | 0 | 0 | 0
    Caregivers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Caregivers: Black or African American | 0 | 0 | 0
    Caregivers: White | 44 | 46 | 90
    Caregivers: More than one race | 0 | 0 | 0
    Caregivers: Unknown or Not Reported | 6 | 7 | 13
Region of Enrollment [Number; unit: participants] — Region of Enrollment for patients only Population: Region of Enrollment for patients only
  participants
    United States: number analyzed (Participants) | 130 | 135 | 265
    United States | 130 | 135 | 265
Region of Enrollment [Number; unit: participants] — Region of enrollment for caregivers only Population: Region of enrollment for caregivers only
  participants
    United States: number analyzed (Participants) | 50 | 53 | 103
    United States | 50 | 53 | 103

OUTCOME MEASURES:

1. Primary Outcome: Mean Patient-centered Communication in Advanced Cancer Score
Description: We audio recorded the first physician visit after the coaching session (for intervention) or after study entry (control).The primary outcome was a composite of 4 pre-specified communication measures: 1. engaging patients in consultations, responding to patients' emotions, informing patients about prognosis and treatment choices and balanced framing of decisions. Coding of the 4 measures was performed by teams of trained university students who were audited continuously and blinded to study hypotheses and group assignment. We transformed each of the 4 component scores to z scores based on the pre-randomization phase sample means (SDs): z = (Raw Score - Pre-randomization Phase Mean)/Pre-randomization Phase SD. The 4-component z-scores were averaged to form the primary outcome. A higher Z score indicates better communication. The maximum possible Z-score ranged from -0.69 to 20.08.
Time Frame: 3 years
Population: This outcome measure was assessed in patients only.
Measure: Mean (Standard Deviation); unit: standardized score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 130 | 135
standardized score on a scale | 0.16 (0.81) | -0.01 (0.66)
Statistical Analysis 1: Comparison: Intervention vs Control; The primary outcome was a composite of 4 prespecified communication measures matched to the goals of communication training, as follows: Active Patient Participation Coding [APPC], Verona VR-CoDES, Prognostic and Treatment Choices [PTCC] Informing subscale, and PTCC Balanced Framing subscale. The 4 measures were z-score transformed and averaged to produce the composite measure; Test type: Superiority; p = 0.05, Mixed Models Analysis; Adjusted mean difference in difference = 0.34, 95% CI 2-sided [0.06 to 0.62] — Models included fixed-effects terms for phase (pre- vs postrandomization), study arm, and the Phase*Arm interaction. Estimated effect is the between-arm difference in adjusted mean difference from prerandomization to postrandomization samples

2. Secondary Outcome: Caregiver Mean Prolonged Grief Symptoms as Measured by PG-13
Description: The prolonged grief (PG-13) instrument was used to measure prolonged grief. The tool is a sum of ten items that measure separation distress, duration of grief, cognitive, emotional, and behavioral symptoms and impairment criterion. The range of the score is 10-50 with higher scores indicating more severe symptoms.
Time Frame: 7 months
Population: This instrument was used with caregivers only.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention: Communication | Control: Usual Care
Number analyzed (Participants) | 48 | 49
units on a scale | 19.3 (5.9) | 20.6 (6.8)
Statistical Analysis 1: Comparison: Intervention: Communication vs Control: Usual Care; Test type: Superiority; p = 0.214, Mixed Models Analysis

3. Secondary Outcome: Aim 1b&c Mean Difference in Reported Expectation of Survival in 2 Years Between Patients and Physicians
Description: Patients and physicians were asked what the likelihood of survival in 2 years would be for the patient. They chose from 0, 10, 25, 50, 75, 90, 100% chance of survival in two years. A value of 0-6 was assigned to each pair of data. 0 indicating no difference in the reported value between patient and physician and 6 indicating the largest difference. For example if the physician said 100% and the patient said 0% the score was 6. The mean scores were reported by arm.
Time Frame: 3 years
Population: This outcome measure was assessed in patients only.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 130 | 135
units on a scale | 2.2 (1.5) | 2.5 (1.6)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.05, Mixed Models Analysis; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.56 to 0.37]

4. Secondary Outcome: Aim 2 Patient Well-being
Description: Original McGill quality of life and the FACT-G assessment tools were used. For the McGill tool scores range from 1 to 10 with higher scores indicating better outcome. For FACT-G scores range from 0 to 4. Higher score means a better outcome. Different parts of the McGill and FACT-G tools were used to create 5 standardized z scores: McGill QOL Scale single item, McGill Psychological Well-Being sub-scale, McGill Existential Well-Being sub-scale, FACT-G Physical Functioning sub-scale and FACT-G Social Functioning sub-scale. Sum of the five standardized z-scores is the Aggregate QOL score. A higher Z score indicates better outcomes. The maximum possible Z-score ranged from -3.54 to 1.24.
Time Frame: 3 years
Population: This outcome measure was assessed in patients only.
Measure: Mean (Standard Deviation); unit: standardized score on a scale
Arm/Group | Intervention: Communication | Control: Usual Care
Number analyzed (Participants) | 130 | 135
standardized score on a scale | -0.01 (0.73) | -0.07 (0.80)

5. Secondary Outcome: Caregiver Mean Overall Mental Health as Measured by the SF-12 Assessment
Description: SF-12 scores are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: 7 months
Population: Sf-12 was given to the caregivers only.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention: Communication | Control: Usual Care
Number analyzed (Participants) | 48 | 49
units on a scale | 48.9 (9.6) | 47.9 (11.5)
Statistical Analysis 1: Comparison: Intervention: Communication vs Control: Usual Care; Test type: Superiority; p = 0.677, Mixed Models Analysis

6. Secondary Outcome: Health Care Utilization- Mean Index Score of Aggressive Care at the End of Life
Description: Patient charts were audited for 3 outcomes : 1) chemotherapy use, 2) aggressive treatments and 3) emergency department or hospital utilization. The total scores ranged from 0-6 with higher scores indicated worse outcomes. The sums of the means for the 3 outcomes were added to provide the total score.
Time Frame: 3 years
Population: Health care utilization was assessed in patients only.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 130 | 135
units on a scale | 0.76 (1.1) | 0.58 (0.9)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.19, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 3 years
Description: There were 91 deaths in the intervention arm for the patients and 1 caregiver death. These were terminally ill patients. Adverse events were not collected for the physicians.
Groups:
- Intervention-patients; Intervention- Caregivers: Oncologists will receive communication training. Patients will be coached to make the most of the oncologist visit.
  Communication training and coaching: Oncologists will receive communication training. Patients will be coached to make the most of the oncologist visit.
- Control-patients; Intervention-caregivers: Patients will receive usual care
Arm/Group | Intervention-patients | Control-patients | Intervention- Caregivers | Intervention-caregivers
All-Cause Mortality (participants affected / at risk) | 91/139 | 96/142 | 1/105 | 0/99
Serious Adverse Events (participants affected / at risk) | 0/139 | 0/142 | 0/105 | 0/99
Other Adverse Events (participants affected / at risk) | 0/139 | 0/142 | 0/105 | 0/99

LIMITATIONS AND CAVEATS:
This was a study of terminally ill patients and all deaths were expected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-02-20): https://cdn.clinicaltrials.gov/large-docs/27/NCT01485627/Prot_000.pdf
  • Statistical Analysis Plan (2016-03-12): https://cdn.clinicaltrials.gov/large-docs/27/NCT01485627/SAP_001.pdf